CLINICAL TRIAL: NCT06492291
Title: A Phase 3, Open-label Extension Study to Evaluate the Safety and Efficacy of MK-0616 in Adults With Hypercholesterolemia
Brief Title: Open-label Extension Study of Enlicitide Decanoate (MK-0616/Enlicitide Oral PCSK9 Inhibitor) in Adults With Hypercholesterolemia (MK-0616-019) CORALreef Extension
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0616-019; 2023-504922-20-00 (Registry Identifier: EU CT); U1111-1290-3950 (Registry Identifier: UTN); jRCT2051240110 (Registry Identifier: jRCT); MK-0616-019 (Other: MSD)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enlicitide Decanoate (Experimental): Participants will receive 20 mg of enlicitide decanoate orally once daily (QD)
  Interventions: Drug: Enlicitide Decanoate

INTERVENTIONS:
Drug: Enlicitide Decanoate — Oral tablet
  Other Names: MK-0616; Enlicitide

SUMMARY:
This is an extension study to evaluate the longer-term safety and efficacy of enlicitide decanoate in adults with hypercholesterolemia who completed either study MK-0616-013 (NCT05952856), study MK-0616-017 (NCT05952869), or study MK-0616-018 (NCT06450366).

ELIGIBILITY:
Inclusion Criteria:

* Has completed an enlicitide decanoate (also known as enlictide and MK-0616) parent study [MK-0616-013 (NCT05952856), MK-0616-017 (NCT05952869), and MK-0616-018 (NCT06450366)] per protocol (including the final assessments/procedures of their parent study)
* Had an overall study intervention compliance ≥80% while participating in their parent study

Exclusion Criteria:

* Has discontinued study intervention in their parent study
* Has an ongoing serious adverse event considered related to study intervention by the investigator in the parent study
* Is planning to begin treatment with a nonstudy protein convertase subtilisin/kexin type 9 inhibitor (PCSK9i) while enrolled in the study
* Is currently participating in an interventional clinical study other than an enlicitide decanoate parent study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2028-10-13 (Estimated); Study Completion 2028-10-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants with one or more adverse events (AEs) | Up to approximately 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study drug due to an AE | Up to approximately 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Mean percent change from baseline of the parent study in LDL-C at Week 8 of this extension study | Baseline of the parent study and Week 8 of this extension study
  The percent change from baseline in LDL-C. Each participant's baseline data from their parent study will be used as baseline data for this analysis.
Mean percent change from baseline of the parent study in non-high-density lipoprotein cholesterol (non-HDL-C) at Week 8 of this Extension Study | Baseline of the parent study and Week 8 of this extension study
  The percent change from baseline in Non-HDL-C. Each participant's baseline data from their parent study will be used as baseline data for this analysis.
Mean percent change from baseline of the parent study in apolipoprotein B (ApoB) at Week 8 of this extension study | Baseline of the parent study and Week 8 of this extension study
  The percent change from baseline in apolipoprotein B. Each participant's baseline data from their parent study will be used as baseline data for this analysis.
Percent change from baseline of the parent study in lipoprotein(a) (Lp[a]) at Week 8 of this extension study | Baseline of the parent study and Week 8 of this extension study
  The percent change from baseline in Lp(a). Each participant's baseline data from their parent study will be used as baseline data for this analysis.
Percentage of participants with LDL-C <70 mg/dL and ≥50% reduction from baseline of the parent study | Baseline in the parent study and up to approximately 3 years in this extension study
  The percentage of participants who have LDL-C <70 mg/dL and ≥50% reduction from baseline at any point during the study. Each participant's baseline data from their parent study will be used as baseline data for this analysis.
Percentage of participants with LDL-C <55 mg/dL and ≥50% reduction from baseline of the parent study | Baseline in the parent study and up to approximately 3 years in this extension study
  The percentage of participants who have LDL-C <55 mg/dL and ≥50% reduction from baseline at any point during the study. Each participant's baseline data from their parent study will be used as baseline data for this analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (222):
- United States (52):
  - Alliance for Multispecialty Research, LLC ( Site 0027), Daphne, Alabama
  - G&L Research ( Site 0035), Foley, Alabama
  - Synexus Clinical Research US, Inc.-Synexus Clinical Research US, Inc - Central Phoenix ( Site 0048), Phoenix, Arizona
  - National Heart Institute-Research ( Site 0029), Beverly Hills, California
  - Clinical Trials Research ( Site 0054), Sacramento, California
  - Velocity Clinical Research, Banning ( Site 0023), San Bernardino, California
  - Emerson Clinical Research Institute ( Site 0017), Washington D.C., District of Columbia
  - Excel Medical Clinical Trials ( Site 0010), Boca Raton, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0037), Doral, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0056), Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach ( Site 0053), Hallandale, Florida
  - Jacksonville Center for Clinical Research ( Site 0025), Jacksonville, Florida
  - South Broward Research ( Site 0012), Miramar, Florida
  - Progressive Medical Research ( Site 0033), Port Orange, Florida
  - Clinical Research Trials of Florida ( Site 0006), Tampa, Florida
  - Clinical Site Partners, LLC dba Flourish Research ( Site 0004), Winter Park, Florida
  - East Coast Institute for Research, LLC ( Site 0020), Macon, Georgia
  - Healthcare Research Network - Chicago ( Site 0051), Flossmoor, Illinois
  - Synexus Clinical Research US - Evansville ( Site 0005), Evansville, Indiana
  - Midwest Institute For Clinical Research ( Site 0052), Indianapolis, Indiana
  - Alliance for Multispecialty Research, LLC ( Site 0001), Lexington, Kentucky
  - L-MARC Research Center ( Site 0011), Louisville, Kentucky
  - Velocity Clinical Research, Covington ( Site 0026), Covington, Louisiana
  - Velocity Clinical Research Rockville ( Site 0022), Rockville, Maryland
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division ( Site 0018), Troy, Michigan
  - Velocity Clinical Research, Gulfport ( Site 0032), Gulfport, Mississippi
  - Healthcare Research Network - St. Louis ( Site 0040), Hazelwood, Missouri
  - Velocity Clinical Research at The Pioneer Heart Institute, Lincoln ( Site 0031), Lincoln, Nebraska
  - Jubilee Clinical Research ( Site 0049), Las Vegas, Nevada
  - AB Clinical Trials ( Site 0002), Las Vegas, Nevada
  - New Mexico Clinical Research & Osteoporosis Center ( Site 0043), Albuquerque, New Mexico
  - Velocity Clinical Research, Syracuse ( Site 0014), East Syracuse, New York
  - Icahn School of Medicine at Mount Sinai-Cardiology ( Site 0042), New York, New York
  - Lillestol Research ( Site 0030), Fargo, North Dakota
  - altoona center for clinical research ( Site 0024), Duncansville, Pennsylvania
  - Cardiology Consultants of Philadelphia Yardley ( Site 0021), Yardley, Pennsylvania
  - Velocity Clinical Research, Anderson ( Site 0015), Anderson, South Carolina
  - Piedmont Research Partners ( Site 0045), Fort Mill, South Carolina
  - Coastal Carolina Research Center ( Site 0055), North Charleston, South Carolina
  - Monument Health Clinical Research, a department of Monument -Monument Health Clinical Research, a d ( Site 0038), Rapid City, South Dakota
  - Holston Medical Group ( Site 0034), Kingsport, Tennessee
  - Alliance for Multispecialty Research, LLC ( Site 0050), Knoxville, Tennessee
  - Velocity Clinical Research, Dallas ( Site 0028), Dallas, Texas
  - Center for Cardiometabolic Disease Prevention/Baylor College of Medicine ( Site 0009), Houston, Texas
  - Clinical Trials of Texas, LLC ( Site 0016), San Antonio, Texas
  - Synexus Clinical Research US, Inc. ( Site 0003), Salt Lake City, Utah
  - Velocity Clinical Research, Salt Lake City ( Site 0041), West Jordan, Utah
  - Manassas Clinical Research Center ( Site 0007), Manassas, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0019), Newport News, Virginia
  - Alliance for Multispecialty Research, LLC ( Site 0008), Norfolk, Virginia
  - National Clinical Research, Inc ( Site 0044), Richmond, Virginia
  - Rainier Clinical Research Center ( Site 0013), Renton, Washington
- Argentina (8):
  - CEDIC ( Site 0603), CABA, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada ( Site 0605), CABA, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0602), Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate ( Site 0604), Zárate, Buenos Aires
  - Fundacion Estudios Clinicos ( Site 0601), Rosario, Santa Fe Province
  - Centro de Investigaciones Metabolicas CINME - Cardiology ( Site 0607), CABA
  - CIPREC ( Site 0600), CABA
  - Fundación Respirar ( Site 0606), CABA
- Australia (2):
  - Royal Prince Alfred Hospital-6West CV Ambulatory Care ( Site 2808), Camperdown, New South Wales
  - Victorian Heart Hospital-Monash Cardiovascular Research Centre (MCRC) ( Site 2803), Clayton, Victoria
- Brazil (3):
  - Universidade Federal Do Ceara ( Site 0702), Fortaleza, Ceará
  - Instituto Dante Pazzanese de Cardiology ( Site 0701), São Paulo, São Paulo
  - Incor - Instituto do Coracao ( Site 0703), São Paulo
- Canada (6):
  - The Medical Arts Health Research Group ( Site 0506), North Vancouver, British Columbia
  - Cambridge Cardiac Care Centre ( Site 0502), Cambridge, Ontario
  - North York Diagnostic and Cardiac Centre ( Site 0505), North York, Ontario
  - Ecogene-21 ( Site 0500), Chicoutimi, Quebec
  - Institut de Cardiologie de Montreal ( Site 0504), Montreal, Quebec
  - Diex Recherche Trois-Rivieres ( Site 0503), Trois-Rivières, Quebec
- Chile (3):
  - Clinical Research Chile SpA ( Site 0800), Valdivia, Los Ríos Region
  - CDIEM ( Site 0801), Providencia, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-CICUC ( Site 0803), Santiago, Region M. de Santiago
- China (18):
  - Beijing Anzhen Hospital, Capital Medical University-Cardiovascular ( Site 6000), Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliate of Capital University ( Site 6003), Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University ( Site 6020), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 6021), Chongqing, Chongqing Municipality
  - Guangdong Provincial People s Hospital ( Site 6004), Guangzhou, Guangdong
  - Zhujiang Hospital ( Site 6029), Guangzhou, Guangdong
  - Huizhou Municipal Central Hospital ( Site 6079), Huizhou, Guangdong
  - The University of Hong Kong-Shenzhen Hospital ( Site 6018), Shenzhen, Guangdong
  - Jingzhou Central Hospital ( Site 6076), Jingzhou, Hubei
  - Wuhan Fourth Hospital ( Site 6056), Wuhan, Hubei
  - Hunan Provincial People's Hospital ( Site 6017), Changsha, Hunan
  - Changzhou Second People's Hospital ( Site 6073), Changzhou, Jiangsu
  - Northern Jiangsu People s Hospital ( Site 6008), Yangzhou, Jiangsu
  - The Third Hospital of Nanchang - Fuhe ( Site 6078), Nanchang, Jiangxi
  - Siping Central People's Hospital ( Site 6011), Siping, Jilin
  - Xianyang Hospital of Yan'an University ( Site 6040), Xianyang, Shaanxi
  - Chengdu Second Municipal People's Hospital ( Site 6032), Chengdu, Sichuan
  - Lishui City People s Hospital ( Site 6002), Lishui, Zhejiang
- Colombia (6):
  - Fundación Centro de Investigación Clínica CIC ( Site 0904), Medellín, Antioquia
  - Ciensalud Ips S A S ( Site 0900), Barranquilla, Atlántico
  - Clinica de la Costa S.A.S. ( Site 0901), Barranquilla, Atlántico
  - Salud SURA Calle 100 ( Site 0905), Bogotá, Cundinamarca
  - Healthy Medical Center S.A.S ( Site 0902), Zipaquirá, Cundinamarca
  - Fundación Valle del Lili ( Site 0903), Cali, Valle del Cauca Department
- Czechia (3):
  - Fakultni Nemocnice u sv. Anny v Brne ( Site 3604), Brno, Brno-mesto
  - Fakultní nemocnice Brno Bohunice-Interni kardiologicka klinika ( Site 3602), Brno, Brno-mesto
  - Institut Klinicke a Experimentalni Mediciny ( Site 3601), Prague, Praha 4
- Meilahden tornisairaala - Meilahti Tower Hospital ( Site 1300), Helsinki, Uusimaa, Finland
- France (3):
  - Hôpital Arnaud de Villeneuve - CHU Montpellier ( Site 5002), Montpellier, Herault
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes ( Site 5004), Saint-Herblain, Loire-Atlantique
  - Hospices Civils de Lyon - Hopital Louis Pradel-Service d'endocrinologie, de diabétologie et des mal ( Site 5000), Bron, Rhone
- Germany (6):
  - Unterfrintroper Hausarztzentrum Klinische Forschung ( Site 1543), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden-Universitätsstudienzentrum für Stoffwechselerkranku ( Site 1510), Dresden, Saxony
  - Hausarzt- und Diabetologische Schwerpunktpraxis Hohenmölsen - Weiβenfels ( Site 1528), Hohenmölsen, Saxony-Anhalt
  - Zentralklinik Bad Berka ( Site 1531), Bad Berka, Thuringia
  - Velocity Clinical Research GmbH Berlin ( Site 1503), Berlin
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin ( Site 1534), Berlin
- Hong Kong (2):
  - Queen Mary Hospital-Medical ( Site 3300), Hksar
  - Prince of Wales Hospital ( Site 3304), Shatin
- Hungary (3):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Belgyógyászati Klinika ( Site 1603), Szeged, Csongrád megye
  - Semmelweis Egyetem-Városmajori Szív- és Érgyógyászati Klinika ( Site 1600), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Belgyógyászati Klinika (Anyagcsere Tanszék) ( Site 1601), Debrecen
- Israel (13):
  - Hillel Yaffe Medical Center ( Site 1731), Hadera
  - Rambam Health Care Campus ( Site 1739), Haifa
  - Rambam Health Care Campus ( Site 1742), Haifa
  - Shaare Zedek Medical Center ( Site 1735), Jerusalem
  - Hadassah Medical Center ( Site 1732), Jerusalem
  - Hadassah Medical Center ( Site 1741), Jerusalem
  - Hadassah Medical Center-Heart Institute ( Site 1734), Jerusalem
  - Meir Medical Center. ( Site 1737), Kfar Saba
  - Rabin Medical Center ( Site 1738), Petah Tikva
  - Rabin Medical Center ( Site 1740), Petah Tikva
  - Sheba Medical Center ( Site 1733), Ramat Gan
  - Clalit Health Services - Sakhnin Community Clinic ( Site 1730), Sakhnin
  - Yitzhak Shamir Medical Center. ( Site 1736), Ẕerifin
- Italy (5):
  - Fondazione Policlinico Tor Vergata ( Site 1809), Rome, Lazio
  - Centro Cardiologico Monzino ( Site 1804), Milan, Milano
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino ( Site 1801), Turin, Piedmont
  - Azienda Ospedaliera Sant'Andrea-Department of Clinical and Molecular Medicine ( Site 1807), Rome, Roma
  - Azienda Ospedaliera Garibaldi ( Site 1810), Catania
- Japan (23):
  - Hirohata Naika Clinic ( Site 3513), Kitakyushu, Fukuoka
  - Nakakinen clinic ( Site 3510), Naka, Ibaraki
  - Noritake Clinic ( Site 3512), Ushiku, Ibaraki
  - National Hospital Organization Kanazawa Medical Center ( Site 3508), Kanazawa, Ishikawa-ken
  - Hirano Medical Clinic ( Site 3522), Morioka, Iwate
  - Shirai Healthcare Clinic Izumichuou ( Site 3527), Sendai, Miyagi
  - Rinku General Medical Center ( Site 3503), Izumisano, Osaka
  - Shiraiwa Medical Clinic ( Site 3514), Kashihara, Osaka
  - Medical Corporation Heishinkai OCROM Clinic ( Site 3501), Suita-shi, Osaka
  - Saitama Medical University Hospital ( Site 3506), Iruma, Saitama
  - Teramoto Medical and Dental Clinic ( Site 3507), Bunkyo-ku, Tokyo
  - Tokyo-Eki Center-building Clinic ( Site 3505), Chuo-ku, Tokyo
  - Fukuwa Clinic ( Site 3504), Chuo-ku, Tokyo
  - Teikyo University Hospital ( Site 3500), Itabashi-ku, Tokyo
  - Kato Clinic of Internal Medicine ( Site 3509), Katsushika-ku, Tokyo
  - Kanno Naika ( Site 3511), Mitaka, Tokyo
  - Sugawara Clinic ( Site 3519), Nerima-ku, Tokyo
  - Shin Clinic ( Site 3517), Ōta-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic ( Site 3502), Shinjuku-ku, Tokyo
  - Medical Corporation Hakuaikai Wellness Tenjin Clinic ( Site 3520), Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital ( Site 3518), Hiroshima
  - Mishuku Hospital ( Site 3524), Tokyo
  - Mitsukoshi Health and Welfare Foundation ( Site 3521), Tokyo
- Mexico (2):
  - Instituto Jalisciense de Investigacion en Diabetes y Obesidad-Endocrinology ( Site 1057), Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador -Unidad de Investigación de Enfermedade ( Site 1071), Mexico City, Mexico City
- Netherlands (4):
  - Radboudumc-internal medicine ( Site 1952), Nijmegen, Gelderland
  - Amsterdam UMC, locatie AMC-Vascular Medicine Clin Trial Unit ( Site 1954), Amsterdam, North Holland
  - Dijklander Ziekenhuis ( Site 1953), Hoorn, North Holland
  - Universitair Medisch Centrum Utrecht-Vascular Medicine Research ( Site 1955), Utrecht
- New Zealand (2):
  - Pacific Clinical Research Network - Rotorua ( Site 2902), Rotorua, Bay of Plenty
  - New Zealand Clinical Research (Christchurch) ( Site 2901), Christchurch, Canterbury
- Norway (2):
  - Nordlandssykehuset ( Site 2041), Bodø, Nordland
  - Oslo Universitetssykehus Aker-Lipidklinikken ( Site 2040), Oslo
- Changi General Hospital ( Site 3211), Singapore, Central Singapore, Singapore
- South Africa (6):
  - IATROS International ( Site 2204), Bloemfontein, Free State
  - Charlotte Maxeke Johannesburg Academic Hospital ( Site 2202), Johannesburg, Gauteng
  - Soweto Clinical Trials Centre ( Site 2203), Soweto, Gauteng
  - TREAD Research ( Site 2201), Cape Town, Western Cape
  - Tiervlei Trial Centre ( Site 2205), Cape Town, Western Cape
  - University of Cape Town (UCT)-Medicine, Division of Lipidology ( Site 2200), Cape Town, Western Cape
- South Korea (15):
  - Wonju Severance Christian Hospital ( Site 3008), Wŏnju, Kang-won-do
  - Chonnam National University Hospital ( Site 3014), Gwangju, Kwangju-Kwangyokshi
  - Seoul National University Bundang Hospital ( Site 3005), Seongnam, Kyonggi-do
  - Ajou University Hospital ( Site 3006), Suwon, Kyonggi-do
  - Chungbuk National University Hospital ( Site 3011), Cheongju-si, North Chungcheong
  - Dong-A University Hospital-Cardiology ( Site 3013), Busan, Pusan-Kwangyokshi
  - Pusan National University Hospital-Internal Medicine ( Site 3012), Busan, Pusan-Kwangyokshi
  - Inje University Haeundae Paik Hospital ( Site 3010), Haeundae-gu, Pusan-Kwangyokshi
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 3003), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 3001), Seoul
  - Kangbuk Samsung Hospital ( Site 3009), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 3002), Seoul
  - Asan Medical Center ( Site 3004), Seoul
  - Samsung Medical Center-cardiology ( Site 3000), Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital-cardiology ( Site 3007), Seoul
- Spain (15):
  - Hospital Universitario Virgen de la Victoria-UGC Endocrinologia y nutricion ( Site 2358), Málaga, Andalusia
  - EBA CENTELLES ( Site 2319), Centelles, Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 2362), Barcelona, Catalonia
  - Hospital de Figueres ( Site 2361), Figueres, Gerona
  - Hospital Abente y Lago ( Site 2356), A Coruña, La Coruna
  - Hospital San Rafael de Coruna ( Site 2363), A Coruña, La Coruna
  - CHUS - Hospital Clinico Universitario-Cardiology - Clinical Research Unit ( Site 2320), Santiago de Compostela, La Coruna
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 2344), Pozuelo de Alarcón, Madrid
  - Hospital Universitario Fundacion ALcorcon-Endocrinologia y Nutrición ( Site 2316), Alcorcón, Madrid, Comunidad de
  - Vithas Hospital Sevilla-Unidad de Salud Metabólica. Diabetes y Obesidad ( Site 2349), Castilleja de la Cuesta, Sevilla
  - Hospital Universitari Sant Joan de Reus ( Site 2329), Reus, Tarragona
  - HOSPITAL CLINICO DE VALENCIA-CARDIOLOGY ( Site 2321), Valencia, Valenciana, Comunitat
  - EAP Sardenya ( Site 2357), Barcelona
  - Hospital Universitario 12 de Octubre-Internal Medicine. Unidad de Ensayos Clínicos ( Site 2311), Madrid
  - Hospital Universitario Virgen Macarena-Cardiology ( Site 2352), Seville
- Taiwan (10):
  - Mackay Memorial Hospital -Tamsui Branch ( Site 3109), New Taipei City, New Taipei
  - Chi Mei Medical Center ( Site 3104), Tainan, Tainan
  - Shin Kong Wu Ho-Su Memorial Hospital ( Site 3110), Taipei City, Taipei
  - Changhua Christian Hospital ( Site 3101), Changhua
  - Chang Gung Memorial Hospital at Kaohsiung ( Site 3102), Kaohsiung City
  - National Cheng Kung University Hospital-Internal Medicine ( Site 3107), Tainan
  - National Taiwan University Hospital ( Site 3100), Taipei
  - Taipei Medical University Hospital ( Site 3108), Taipei
  - Taipei Veterans General Hospital ( Site 3106), Taipei
  - Chang Gung Medical Foundation-Linkou Branch ( Site 3105), Taoyuan District
- Turkey (Türkiye) (6):
  - Ege Universitesi Hastanesi-Cardilogy Department ( Site 2502), Bornova, İzmir
  - Hacettepe Universite Hastaneleri ( Site 2500), Ankara
  - Ankara Bilkent Şehir Hastanesi-cardiology ( Site 2501), Ankara
  - Eskisehir Osmangazi University-Cardiology ( Site 2510), Eskişehir
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri ( Site 2522), Kayseri
  - Kocaeli Üniversitesi-Cardiology ( Site 2516), Kocaeli
- United Kingdom (2):
  - Barts Health NHS Trust-William Harvey Clinical Research Centre ( Site 4001), London, England
  - Royal Free Hospital ( Site 4000), London, England

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26122&tenant=MT_MSD_9011